CLINICAL TRIAL: NCT06242353
Title: Coagulopathy in Childhood Acute Lymphoblastic Leukaemia, Underlying Mechanisms and Ways to Optimise Treatment
Brief Title: Coagulopathy in Childhood Acute Lymphoblastic Leukaemia
Acronym: CoagCALL
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Mats Heyman, Associate Professor, Consultant, Karolinska University Hospital
Other Study IDs: K2021-5396
Record Dates: First submitted 2023-10-03; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Acute Lymphoblastic Leukemia; Thrombosis; Bleeding; Hemostatic Disorder
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Thrombosis; Hemorrhage; Hemostatic Disorders | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coagulopathy parameters — Standard coagulation tests: APT (Activated Partial Thromboplastin Time), PT/INR (Prothrombin Time Test), Protein-C, Protein-S, Fibrinogen, Antithrombin, D-dimers.
  Global haemostasis assays: CAT (Calibrated Automated Thrombogram), OHP (Overall Haemostatic Potential), Fibrin clot turbidity assay, microparticle detection by flow cytometry, scanning electron microscopy.
  Protein expression profile (mass spectroscopy)
  Ultrasound of catheterised neck veins to detect clots
  Other Names: Ultrasound

SUMMARY:
The goal of this study is to investigate the hemostatic balance in children with acute lymphoblastic leukaemia (ALL) treated according to the ALLTogether1 protocol with focus on the early treatment period including concomitant use of steroids and asparaginase.

The investigators aim to determine if complement proteins or microparticles can be used as clinically relevant predictive or diagnostic biomarkers for thrombosis and if global hemostatic assays can predict bleeding or thrombosis. Characterization of proteins connected to hemostasis before and during ALL treatment may provide pathophysiological insights regarding ALL- and treatment related coagulopathy. The ultimate goal of the study is to minimize the morbidity and mortality related to thrombosis and bleeding complications in children with ALL.

Several pediatric oncology centers in Sweden will be participating in this study, which will enroll approximately 100 pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Lymphoblastic Leukaemia (ALL) in Sweden
* Age 1-17.99 years at diagnosis
* Planned/Initiated treatment for ALL according to the ALLTogether1 protocol
* Signed informed consent from parents and patients (from 12 years - voluntary if <15 years)

Exclusion Criteria:

* Other underlying diseases which according to examiner's clinical assessment may increase the risk of bleeding or thrombosis and which are expected to lead to adaption of the therapy protocol for ALL (e g APS, moderate/severe v Willebrand disease, haemophilia)
* Patient not treated according to the ALLTogether1 protocol (including patients with BCR::ABL1, mixed phenotype acute leukaemia - MPAL)

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients fulfilling inclusion criteria and without exclusion criteria diagnosed at participating centres (Stockholm, Uppsala, Linköping, Lund).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Coagulation events (thrombosis and/or bleeding) in early phases of treatment for childhood ALL according to the ALLTogether1 therapy protocol | From diagnosis until the start of the subsequent phase of therapy (day 0 to 106 in protocol therapy)
  Incidence of coagulation events during the induction and consolidation phases (first 106 days of ALL-therapy)

SECONDARY OUTCOMES:
Laboratory abnormalities indicating a risk of haemostatic events in the early phases of childhood ALL therapy | From diagnosis until the start of the subsequent phase of therapy (day 0 to 106 in protocol therapy)
  Incidence of laboratory abnormalities during the induction and consolidation phases (first 106 days of ALL-therapy)
Sub-clinical catheter-related thrombosis (central vein catheters) during the early phases of childhood ALL therapy | At the end of induction (protocol day 29 +/- 3 days)
  Thrombosis detected by ultrasound screening of catheterised neck veins

IPD SHARING:
Plan to Share IPD: No
When study has been completed and published, IPD may be shared with other researchers on collaborative basis, provided that data protection for study subjects can be ensured and that no violation of data-protection legislation will occur.